CLINICAL TRIAL: NCT04152382
Title: A Multiple-Dose, Randomized, Placebo-Controlled, Study of LY3462817 or LY3509754 in Patients With Psoriasis
Brief Title: A Safety Study of LY3462817 and LY3509754 in Participants With Psoriasis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to liver findings
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17218; J1A-MC-KDAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-11-04; First posted 2019-11-05 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY3462817 - Intravenous (IV) (Experimental): LY3462817 administered as IV infusions.
  Interventions: Drug: LY3462817 - IV
- Placebo - IV (Placebo Comparator): Placebo administered as IV infusions.
  Interventions: Drug: Placebo - IV
- LY3462817 - Subcutaneous (SC) (Experimental): LY3462817 administered as SC injections. (SC administration is discretionary/optional.)
  Interventions: Drug: LY3462817 - SC
- Placebo - SC (Placebo Comparator): Placebo administered as SC injections. (SC administration is discretionary/optional.)
  Interventions: Drug: Placebo - SC
- LY3509754 (Experimental): LY3509754 administered orally.
  Interventions: Drug: LY3509754
- Placebo (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3462817 - IV — Administered IV
  Arms: LY3462817 - Intravenous (IV)
Drug: LY3462817 - SC — Administered SC
  Arms: LY3462817 - Subcutaneous (SC)
Drug: Placebo - IV — Administered IV
  Arms: Placebo - IV
Drug: Placebo - SC — Administered SC
  Arms: Placebo - SC
Drug: LY3509754 — Administered orally.
  Arms: LY3509754
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
This study is being conducted to determine how safe and how well tolerated LY3462817 is when given to participants with psoriasis. Blood tests will be done to check how much LY3462817 is in the bloodstream and how long the body takes to get rid of it. The study will last up to one year and one month for each participant. As part of protocol addendum, this study is additionally evaluating the safety and tolerability of LY3509754 in participants with psoriasis. Blood tests will be done to check how much LY3509754 is in the bloodstream and how long the body takes to get rid of it. The addendum will last up to 12 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been diagnosed with psoriasis for at least 6 months
* Participants must have active psoriasis plaques
* Participants must be willing and able to have skin biopsies (small samples of skin removed for testing)

Exclusion Criteria:

* Participants must not have received certain medications for psoriasis that are applied to the skin within 14 days prior to baseline (Day 1)
* Participants must not have received certain oral or injectable medications or light therapy for psoriasis within 4 weeks prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to LY3462817 and LY3509754 | Baseline through Final Follow-up (up to Week 52 for LY3462817 & up to Week 16 for LY3509754)
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Average Concentration (Cave) of LY3462817 and LY3509754 | Baseline through Final Follow-up (up to Week 52 for LY3462817 & up to Week 16 for LY3509754)
  PK: Cave of LY3462817 and LY3509754

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (10):
  - Dermatology Associates - Los Angeles, Los Angeles, California
  - Miami Dermatology and Laser Research, Miami, Florida
  - Advanced Pharma Clinical Research, Miami, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Avita Clinical Research, Tampa, Florida
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - DermDox Centers for Dermatology, Hazleton, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
- Canada (3):
  - Simcoderm Medical & Surgical Dermatology Centre, Barrie, Ontario
  - Skin Health, Cobourg, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Safety Study of LY3462817 in Participants With Psoriasis — https://trials.lillytrialguide.com/en-US/trial/azmsPbmvZOOmiS1aMi7nO